CLINICAL TRIAL: NCT04286893
Title: Improved Heart Rate Variability, Inflammation Markers and Endothelial Function After Transcatheter Aortic Valve Implantation
Brief Title: Improved HRV, Inflammation Markers and Endothelial Function After TAVI
Acronym: bTAVI
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Luka Vitez, Luka Vitez, MD, cardiology resident, University Medical Centre Ljubljana
Other Study IDs: UKCLbTAVI
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Severe Aortic Stenosis; TAVI
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood withdrawal for endothelial inflammation markers detection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVI group: Consecutive patients undergoing TAVI
  Interventions: Diagnostic Test: Flow mediated vasodilatation; Diagnostic Test: High resolution ECG; Diagnostic Test: Blood withdrawal

INTERVENTIONS:
Diagnostic Test: Flow mediated vasodilatation — Measurement of brachial artery diameter change before and after limb ischaemia.
Diagnostic Test: High resolution ECG — Measurement HRV using high resolution ECG
Diagnostic Test: Blood withdrawal — Measurement of endothelial inflammation markers

SUMMARY:
Severe aortic valve stenosis is known to affect heart haemodynamics, endothelial function and body inflammation markers. Our aim is to investigate the weather transcatheter aortic valve implantation in patients with severe aortic stenosis affects heart rate variability, inflammation markers and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* TAVI

Exclusion Criteria:

* stage V chronic kidney disease
* active malignancies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients eligible for transfemoral transcatheter aortic valve implantation
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change of heart rate variability | 3 to 6 months after TAVI
  Change of heart rate variability (HRV) estimated with digital high resolution ECG recording
Change of laboratory value of endothelial inflammation markers | 3 to 6 months after TAVI
  Laboratory determined numerical changes in endothelial inflammation markers
Change of flow-mediated filatation (FMD) of the brachial artery | 3 to 6 months after TAVI
  % flow-mediated dilatation

CONTACTS AND LOCATIONS:
Overall Officials: Borut Jug, PhD, Study Director — University Medical Centre Ljubljana
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Horn P, Stern D, Veulemans V, Heiss C, Zeus T, Merx MW, Kelm M, Westenfeld R. Improved endothelial function and decreased levels of endothelium-derived microparticles after transcatheter aortic valve implantation. EuroIntervention. 2015 Apr;10(12):1456-63. doi: 10.4244/EIJY14M10_02. PMID 25287265
- [Derived] Vitez L, Starc V, Jug B, Bunc M. Improved Endothelial and Autonomic Function after Transcatheter Aortic Valve Implantation. Rev Cardiovasc Med. 2023 May 8;24(5):140. doi: 10.31083/j.rcm2405140. eCollection 2023 May. PMID 39076751